CLINICAL TRIAL: NCT00303966
Title: A Phase II Study of BAY 43-9006 in Relapsed Chronic Lymphocytic Leukemia
Brief Title: Sorafenib in Treating Patients With Relapsed Chronic Lymphocytic Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02688; 14194B; UCCRC-14194B; NCI-7071; CDR0000462339; N01CM62201 (NIH)
Record Dates: First submitted 2006-03-15; First posted 2006-03-17 (Estimated); Results first posted 2014-04-10 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-01

CONDITIONS: Refractory Chronic Lymphocytic Leukemia; Stage I Chronic Lymphocytic Leukemia; Stage II Chronic Lymphocytic Leukemia; Stage III Chronic Lymphocytic Leukemia; Stage IV Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Sorafenib

ARMS (1):
- Treatment (sorafenib tosylate) (Experimental): Patients receive oral sorafenib twice daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: sorafenib tosylate

INTERVENTIONS:
Drug: sorafenib tosylate — Given orally
  Other Names: BAY 43-9006; BAY 43-9006 Tosylate Salt; BAY 54-9085; Nexavar; SFN

SUMMARY:
Sorafenib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the cancer. This phase II trial is studying how well sorafenib works in treating patients with relapsed chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the objective response rate in patients with recurrent chronic lymphocytic leukemia (CLL) treated with sorafenib.

II. Determine the toxicity in patients treated with sorafenib.

SECONDARY OBJECTIVES:

I. Correlate bone marrow angiogenesis, CLL tumor cell expression of vascular endothelial growth factor (VEGF), VEGF receptors (flt-1, KDR, flt-4 and neuropilin-1), basic fibroblast growth factor, and plasma interleukin-8 levels with response.

OUTLINE: This is a multicenter study.

Patients receive oral sorafenib twice daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: Approximately 40 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed chronic lymphocytic leukemia (CLL) by NCI-WG immunophenotype and blood criteria

  * Documentation of current or prior peripheral blood (PB) or bone marrow (BM) immunophenotype compatible with CLL

    * Patients who currently do not have > 5,000/mm³ absolute lymphocytosis are eligible if they have previously met PB lymphocytosis criteria and have a current immunophenotype documenting monoclonal B lymphocytosis morphologically and immunophenotypically compatible with CLL
* Intermediate-risk (Rai stage I or II) or high-risk (Rai stage III or IV) disease, including any of the following:

  * Rai stage I disease with lymphocytosis and enlarged nodes
  * Rai stage II disease with lymphocytosis plus splenomegaly and/or hepatomegaly (nodes positive or negative)
  * Rai stage III disease with lymphocytosis plus anemia
  * Rai stage IV disease with lymphocytosis and thrombocytopenia
* Must require treatment with active disease, experiencing disease related symptoms, or having deterioration of blood counts, meeting ≥ 1 of the following criteria:

  * Presence of ≥ 1 of the following disease-related symptoms:

    * Weight loss > 10% within the past 6 months
    * Extreme fatigue (i.e., ECOG performance status 2: cannot work or unable to perform usual activities)
    * Fever > 100.5°F for 2 weeks without evidence of infection
    * Night sweats without evidence of infection
  * Evidence of progressive marrow failure, as manifested by worsening of anemia (hemoglobin < 10 g/dL), thrombocytopenia (platelet count < 100,000/mm³), and/or neutropenia (neutrophil count < 2,000/mm³)
  * Massive (i.e., > 6 cm below left costal margin) or progressive splenomegaly or discomfort from splenomegaly
  * Massive nodes or clusters (i.e., > 10 cm in longest diameter), progressive adenopathy, or discomfort from lymphadenopathy
  * Deterioration of blood counts and/or progressive lymphocytosis, with an increase of ≥ 10% documented over a 2-month period OR an anticipated doubling time < 6 months
* Relapsed disease

  * Must receive at least 1, but no more than 3, prior chemotherapy regimens with any cytotoxic agent or antibody therapy

    * No fludarabine refractory disease

      * Responded to prior fludarabine without relapse or disease progression for at least 6 months
* Patients with a history of Coombs-positive hemolytic anemia are eligible provided recovery from treatment of hemolysis and off steroids
* No stage 0 CLL
* No known CNS involvement
* Life expectancy > 6 months
* ECOG performance status 0-2 OR Karnofsky performance status 70-100%
* Absolute neutrophil count ≥ 1,000/mm³
* Platelets ≥ 30,000/mm³
* Bilirubin ≤ 2 mg/dL
* AST/ALT ≤ 2.5 times upper limit of normal (ULN)
* Creatinine ≤ 1.5 times ULN OR creatinine clearance ≥ 60 mL/min (for patients with creatinine levels above normal)
* No currently active second malignancy
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patient must use effective contraception prior to and during study participation
* No uncontrolled hypertension, defined as blood pressure (BP) > 150/100 mm Hg on 2 different measurements at least 1 day apart with either systolic or diastolic number meeting this definition

  * Patients may later enter the study, if they have achieved stable BP (i.e., < 140/90 mm Hg) on a regimen of ≤ 2 drugs after 6-8 weeks of therapy
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to sorafenib
* No uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situations that would limit compliance with the study requirements
* No active infection requiring systemic antibiotics
* No evidence of bleeding diathesis
* No evidence of bowel perforation or obstruction risk
* No swallowing dysfunction leading to difficulty taking the study drug
* See Disease Characteristics
* Recovered from prior therapy
* At least 2 weeks since prior antibiotic therapy
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin C) or radiotherapy
* At least 12 weeks since prior monoclonal antibody
* Concurrent warfarin for anticoagulation allowed provided all of the following are met:

  * On a stable therapeutic dose
  * INR ≤ 3
  * No active bleeding or pathological condition that carries high-risk of bleeding
* No prior MAPK signaling inhibitor agents or anti-angiogenesis agents
* No concurrent combination anti-retroviral therapy for HIV-positive patients
* No concurrent cytochrome P450 enzyme-inducing antiepileptic drugs (phenytoin, carbamazepine, or phenobarbital), rifampin, or Hypericum perforatum (St. John's wort)
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2005-11; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Stock, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (1):
- University of Chicago Comprehensive Cancer Center, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Sorafenib Tosylate)
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Sorafenib Tosylate)
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Objective response is defined as a complete (CR) or partial (PR) remission. Complete remission is defined as no evidence of chronic lymphocytic leukemia (CLL) in marrow with normal hematopoiesis and no palpable lymphadenopathy. Partial remission is defined as improvement in blood counts from baseline with >50% reduction in lymph nodes on examination. These are definitions from the CLL International Working Group (IWG).
Time Frame: Up to week 25
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Sorafenib Tosylate)
Number analyzed (Participants) | 5
percentage of participants | 0 [0 to 52]

2. Primary Outcome: Time to Disease Progression
Description: Time to disease progression will be defined as the time from treatment start until disease progression and will be evaluated using the Kaplan-Meier estimator. Those who do not progress will be censored at the time that they were last known to be progression free.
Time Frame: Up to 5.5 years
Population: Study terminated early and only 5 patients were enrolled.
Measure: Median (Standard Error); unit: months
Arm/Group | Treatment (Sorafenib Tosylate)
Number analyzed (Participants) | 5
months | 4.6 (1.2)

3. Primary Outcome: Overall Survival
Description: Overall survival will be defined as time from the start of treatment until death from any cause and will be evaluated using the Kaplan-Meier estimator.
Time Frame: Up to 5.5 years
Population: Study terminated early and only 5 patients were enrolled.
Measure: Median (Standard Error); unit: months
Arm/Group | Treatment (Sorafenib Tosylate)
Number analyzed (Participants) | 5
months | 32.8 (10.5)

4. Secondary Outcome: Changes in Mean Microvessel Density From Baseline to Week 25
Description: Mean microvessel density will serve as a marker of angiogenesis (other markers includes hot spot density). Will be examined using random-effects linear models.
Time Frame: Baseline and week 25
Population: Study terminated early with only 5 patients. Data wasn't collected for this outcome.
Arm/Group | Treatment (Sorafenib Tosylate)
Number analyzed (Participants) | 0

5. Secondary Outcome: Changes in Vascular Endothelial Growth Factor (VEGF) From Baseline to Week 25
Description: Changes in VEGF levels (post-pretreatment) will be assessed. A negative value indicates a decrease with treatment.
Time Frame: Baseline and week 25
Population: Study terminated early after enrolling only 5 patients. Data wasn't collected for this outcome.
Arm/Group | Treatment (Sorafenib Tosylate)
Number analyzed (Participants) | 0

6. Secondary Outcome: Changes in Plasma Level of Interleukin-8 (IL-8) From Baseline to Week 25
Description: The change (post-pretreatment) will be calculated and tested using a paired t test. A negative value indicates a decrease with treatment.
Time Frame: Baseline and week 25
Population: Study terminated early and enrolled only 5 patients. Data wasn't collected for this outcome.
Arm/Group | Treatment (Sorafenib Tosylate)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: up to 6 months
Description: Grade 3 or higher adverse events are reported.
Arm/Group | Treatment (Sorafenib Tosylate)
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Sorafenib Tosylate) (N=5)
Cholecystitis (Hepatobiliary disorders) | 1
Lung infection (Infections and infestations) | 1
Platelet count decreased (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Sorafenib Tosylate) (N=5)
Anemia (Blood and lymphatic system disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Fatigue (General disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1

LIMITATIONS AND CAVEATS:
Early termination leading to small number of subjects

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less